CLINICAL TRIAL: NCT00599716
Title: A Phase 3, Multicenter, Randomized, Double-Masked Study of Safety and Efficacy of Vismed® in Dry Eye Syndrome
Brief Title: Safety and Efficacy Assessment of Vismed® (Sodium Hyaluronate) for the Treatment of Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lantibio (Industry)
Collaborators: River Plate Biotechnology, Inc. (Industry); Rx Development Resources, LLC (Unknown)
Responsible Party: Terry W. Laliberte/Director of Development, River Plate Biotechnology, Inc./Lantibio, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP-001
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Dry Eye Disease
Keywords: dry eye syndrome; dry eye disease; Vismed; dry eye; sodium hyaluronate; hyaluronic acid
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): study drug
  Interventions: Drug: sodium hyaluronate
- 2 (Placebo Comparator): vehicle control
  Interventions: Drug: vehicle

INTERVENTIONS:
Drug: sodium hyaluronate — a sterile, unpreserved eye drop containing sodium hyaluronate in a proprietary formulation to be administered by ocular instillation
  Other Names: Vismed®; hyaluronic acid
  Arms: 1
Drug: vehicle — identical to proprietary formulation of active eye drop but without active ingredient, sodium hyaluronate
  Arms: 2

SUMMARY:
The study is designed to assess the safety and efficacy of Vismed®, a special eye drop containing sodium hyaluronate, in the treatment of dry eye syndrome. Vismed® is being compared to another eye drop, identical in composition except that it does not contain the active ingredient, sodium hyaluronate. This eye drop is designed as the "vehicle." Some subjects are to receive Vismed® treatment, while others are to receive the vehicle; the assignment of subjects to receive either Vismed or vehicle is to be random. The two-week treatment phase is followed by a one week follow-up period to evaluate safety of Vismed®.

DETAILED DESCRIPTION:
VISMED® is currently marketed in Europe under the CE mark as a viscoelastic lubricant eye drop. The proprietary formulation contains a highly purified specific fraction of sodium hyaluronate. Sodium hyaluronate is a natural polymer which is also present in the structures of the human eye. Its main physical characteristic is viscoelasticity. This means that VISMED® has a high viscosity between blinks and a low viscosity during blinking ensuring efficient coating of the surface of the eye. It is believed that this protective coating of the surface of the eye helps prevent dryness and irritation. Sodium hyaluronate also possesses mucoadhesive properties and the ability to entrap water, thus resembling tear mucus glycoprotein. This, together with the coating properties of sodium hyaluronate, results in an increased pre-corneal residence time and tear film break-up time (BUT) and therefore longer lubrication of the eye surface. VISMED® is completely free of preservatives. As a result, it is non-irritating to ocular tissues and can be used frequently and for extended periods without harming the surface of the eye (e.g. without causing superficial punctate keratitis). Some preservatives are known to cause toxic or allergic reactions, the symptoms of which include stinging, burning and redness of the eyes. To further maximize patient comfort, the pH of VISMED® is adjusted to 7.3, similar to that of the natural tear film.

Hydrogels of sodium hyaluronate have been used for many years in ophthalmic surgery in Europe and the U.S. to maintain the shape of the eye, to cover surgical instruments and to protect the corneal endothelium from damage. They have unique physical properties that make them ideal for use in the treatment of Dry Eye Syndrome. Therefore, VISMED® represents a new class of compound in development for the treatment of dry eye in the US, offering lubricant properties which can alleviate the discomfort and reverse ocular damage caused by dry eye syndrome.

This study is being conducted to supplement the body of knowledge gained from studies conducted in Europe and regulatory approvals granted there to formalize the safety and efficacy of Vismed® to meet FDA requirements for a New Drug Application to market the product in the US.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18 years and over.
* Subjects should have at least a 3-month documented history of dry eye in both eyes diagnosed as dry eye syndrome, keratoconjunctivitis sicca (KCS), or due to Sjögren syndrome (immune exocrinopathy).
* Subjects must agree to discontinue all artificial tears from Screening through the duration of the treatment period (Screening to Day 14).
* Subjects who have taken Restasis® are eligible for inclusion if they have not used Restasis® during the 4 weeks prior to Screening.
* Subjects must discontinue lens wear one week before Screening and agree not to wear contact lenses during the entire study.
* Subjects must provide signed informed consent prior to participation in any study-related procedures.

Exclusion Criteria:

* Pregnancy or lactation.
* Females of childbearing potential who are not using systemic contraception, are not postmenopausal (≥ 1 year), or are not surgically sterilized.
* Ocular surgery (of any type, including laser surgery) or ocular trauma within the 4 months prior to Screening.
* Other diseases or characteristics judged by the investigator to be incompatible with the assessments needed in this study or with reliable instillation of the study medication.
* Any active inflammation of the eye not due to KCS (eg, iritis, scleritis, etc.).
* Participation in any other clinical trial within 30 days prior to Screening.
* Prior participation in a previous clinical trial of Vismed®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
staining of the cornea and conjunctiva | Day 7
symptom frequency score | Day 7

SECONDARY OUTCOMES:
staining of the cornea and conjunctiva | Day 14
symptom frequency score | Day 14
Quality of Life assessment | Day 7 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vogel, MD, Study Chair — Rx Development Resources, LLC; Terry Laliberte, BS, Study Director — River Plate Biotechnology, Inc.; Charles (Andy) Kirby, MD, Principal Investigator — Chattanooga Eye Institute, Chattanooga, TN; Mark Abrams, MD, Principal Investigator — Abrams Eye Center, Cleveland, OH
Locations (10):
- United States (10):
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Center for Excellence in Eye Care, Miami, Florida
  - East Florida Eye Institutue, Stuart, Florida
  - Abrams Eye Center, Stuart, Florida
  - International Eye Center, Tampa, Florida
  - American Eye Institute, New Albany, Indiana
  - Comprehensive Eye Care, Washington, Missouri
  - Charlotte Eye, Ear, Nose and Throat, Charlotte, North Carolina
  - Ophthalmic Research & Clinical Studies, Moon Twp, Pennsylvania
  - Chattanooga Eye Institute, Chattanooga, Tennessee